CLINICAL TRIAL: NCT04896593
Title: Mobile Technology for Reducing and Preventing Adolescent Suicide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hartford Hospital (Other)
Collaborators: Oui Therapeutics, Inc. (Industry); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HHC-2020-0363; R43MH125691 (NIH)
Record Dates: First submitted 2021-05-14; First posted 2021-05-21 (Actual); Results first posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Suicide, Attempted; Suicidal Ideation
MeSH Terms: conditions — Suicide, Attempted; Suicidal Ideation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Smartphone app teaching suicide prevention skills.
  Interventions: Behavioral: Smartphone App

INTERVENTIONS:
Behavioral: Smartphone App — Smartphone app teaching suicide prevention skills.

SUMMARY:
This single-group open-label trial will evaluate the feasibility and preliminary efficacy of a suicide prevention mobile application when used as an adjunct to usual care in adolescents.

DETAILED DESCRIPTION:
This study will enroll 20 adolescent (age 13-17) inpatients at elevated risk for suicide. Participants will download the app onto their phones during their inpatient stay and will complete a single therapy session involving psychoeducation and crisis response planning. Participants will be encouraged to use the app on their own in addition to their usual outpatient services to learn and practice suicide prevention skills. Participants and their parents will be interviewed 1, 4, 8, 12, and 16 weeks after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient psychiatric patients who have attempted suicide (lifetime) or have documented suicide ideation and a plan to harm themselves at admission
* Understand written and spoken English
* Own an iPhone with iOS 11 or higher, or Android with OS 8.1 or higher
* Willing and able to complete enrollment procedures
* Parent/guardian (and youth) able to understand the nature of the study and provide written informed consent (assent for youth)
* Willing to agree to release of information to their parent/guardian and providers when clinically indicated.
* Discharge plan includes aftercare within the Hartford HealthCare system (to facilitate coordination of care during follow up)

Exclusion Criteria:

* Patients with active psychosis
* Patients experiencing substance withdrawal
* Currently enrolled in other treatment studies for the symptoms and behaviors targeted
* Patient unwilling or unable to wear mask during in-person study procedures
* Patients who, in the judgment of the investigator, would have an unfavorable risk/benefit profile with respect to the Smartphone App.
* Any other psychiatric or medical condition (e.g., intellectual disability) or custody arrangement that in the investigator's opinion would preclude informed consent/assent or participation in the trial.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Tolin, Ph.D., Principal Investigator — Institute of Living/Hartford Hospital
Locations (1):
- Institute of Living/Hartford Hospital, Hartford, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention
Started | 22
Completed | 17
Not Completed | 5
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 1
Not completed — Did not complete onboarding | 2

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.8182 (1.2587)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 16
  Gender: Trans male | 2
  Gender: Nonbinary/Genderfluid | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 12
  More than one race | 1
  Unknown or Not Reported | 5
Baseline SIQ [Mean (Standard Deviation); unit: units on a scale] — Population: 2 participants consented but dropped from the study prior to receiving the intervention (app). They were not included in the outcome analysis.
  units on a scale
    number analyzed (Participants) | 20
    (all) | 54.700 (18.966)

OUTCOME MEASURES:

1. Primary Outcome: App Usability 1 Week
Description: The System Usability Scale (SUS) contains 10 items assessing the usability of digital technology. Items are rated from 1 to 5 with higher numbers representing stronger agreement with usability statements. Scores can range from 0 to 100, with higher scores reflecting better outcomes, meaning increased usability of the technology. The mean and standard deviation for the SUS will be reported utilizing all available data.
Time Frame: 1 week post discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 19
score on a scale | 83.948 (10.046)

2. Primary Outcome: App Usability 4 Weeks
Description: as for outcome 1
Time Frame: 4 weeks post discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 16
score on a scale | 86.875 (9.060)

3. Primary Outcome: App Usability 8 Weeks
Description: as for outcome 1
Time Frame: 8 weeks post discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 15
score on a scale | 85.500 (9.171)

4. Primary Outcome: App Usability 12 Weeks
Description: as for outcome 1
Time Frame: 12 weeks post discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 15
score on a scale | 86.833 (10.457)

5. Primary Outcome: App Usability 16 Weeks
Description: as for outcome 1
Time Frame: 16 weeks post discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 16
score on a scale | 85.625 (8.827)

6. Secondary Outcome: Suicidal Ideation Baseline
Description: The SIQ Jr is a 15-item measure assesses suicidal thoughts on a 7-point scale, with possible total scores ranging from 0-90). Higher scores indicate more severe suicidal ideation. Means and standard deviations will be reported utilizing all available data.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 20
score on a scale | 54.700 (18.966)

7. Secondary Outcome: Suicidal Ideation 1 Week
Description: as for outcome 6
Time Frame: 1 Week post discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 19
score on a scale | 43.421 (12.048)

8. Secondary Outcome: Suicidal Ideation 4 Weeks
Description: as for outcome 6
Time Frame: 4 Weeks post discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 16
score on a scale | 27.125 (15.165)

9. Secondary Outcome: Suicidal Ideation 8 Weeks
Description: as for outcome 6
Time Frame: 8 Weeks post discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 15
score on a scale | 25.200 (18.033)

10. Secondary Outcome: Suicidal Ideation 12 Weeks
Description: as for outcome 6
Time Frame: 12 Weeks post discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 15
score on a scale | 26.867 (19.375)

11. Secondary Outcome: Suicidal Ideation 16 Weeks
Description: as for outcome 6
Time Frame: 16 Weeks post discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 16
score on a scale | 26.625 (16.045)

ADVERSE EVENTS:
Time Frame: From study enrollment through 16 weeks post-discharge assessment.
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 9/22
Other Adverse Events (participants affected / at risk) | 19/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=22)
Suicide attempt (Psychiatric disorders) | 4 (4)
Inpatient hospitalization (Psychiatric disorders) | 5 (7)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=22)
Headaches (General disorders) | 1 (1)
Increase in anger (Psychiatric disorders) | 1 (1)
Increase in SIQ-Jr total score above threshold (Psychiatric disorders) | 3 (3) — Increase in SIQ-Jr total score above reliable change threshold
Increased fatigue in swimming (Psychiatric disorders) | 1 (1)
Sinus issue (General disorders) | 1 (1)
Feeling more down (Psychiatric disorders) | 1 (1) — Feeling more down due to increased swim and school demands
Weight gain (General disorders) | 1 (1) — 10lb weight gain at the end of swim season
Medication side effects (Psychiatric disorders) | 1 (1) — Side effects after stopped taking psychiatric medications
Increased mania (Psychiatric disorders) | 1 (1) — Increased mania, frequently leaving house against parental wishes, discontinued psychiatric medications
Sexual assault (Social circumstances) | 1 (1) — Reported sexual assault to police and study IE
Thoughts of self-harm (Psychiatric disorders) | 2 (2)
ER and Urgent Care visits for migraines and vomiting. (General disorders) | 1 (1) — Increased migraines and anxiety, vomiting due to migraines. Having hard time going to school and seeing friends. Went to the ER 3 times and Urgent Care 2 times, not admitted to hospital due to migraines/vomiting
ER visit for dizziness and not eating or drinking (General disorders) | 1 (1) — Transferred from psychiatric inpatient to ER for dizziness and not eating or drinking
COVID-19+ (General disorders) | 1 (1)
ER visit for vomiting (General disorders) | 1 (1)
Increased stress, DCF involvement (Psychiatric disorders) | 1 (1) — Increased stress, patient escorted home after spending the night outside of the home. DCF involved afterwards.
ER visit due to allergic reaction (Immune system disorders) | 1 (1) — Accidental ingestion of nuts (has severe nut allergy), used epi pen. Went to ER and given steroid and Pepcid before discharged. No hospitalization.
Viral respiratory infection (Infections and infestations) | 1 (1) — Not COVID/strep
Passive suicidal ideation, feeling more down (Psychiatric disorders) | 1 (1)
ER visit for suicidal ideation (Psychiatric disorders) | 1 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The principal investigator was designated by the sponsor to be the party responsible for conducting the trial and has the right to publish the results of the trial with approval from the sponsor.

DOCUMENTS (3):
  • Study Protocol (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/93/NCT04896593/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-14): https://cdn.clinicaltrials.gov/large-docs/93/NCT04896593/SAP_001.pdf
  • Informed Consent Form (2021-05-24): https://cdn.clinicaltrials.gov/large-docs/93/NCT04896593/ICF_002.pdf